CLINICAL TRIAL: NCT03630848
Title: Protein Concentration and Human Embryo Development
Brief Title: Effect of Protein Concentration on Human Embryo Development
Acronym: PCHED
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ibn Sina Hospital (Other Government)
Collaborators: Banon IVF Center Assiut, Egypt (Other)
Responsible Party: Principal Investigator, Muhammad Fawzy, ivF Lab Director, Ibn Sina Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: IbnSina IVFCenter-Protein
Record Dates: First submitted 2018-08-10; First posted 2018-08-15 (Actual); Last update posted 2020-06-11 (Actual); Status verified 2020-06

CONDITIONS: Human Embryo Culture

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 10 mg/ml protein concentration in Embryo Culture Media (Experimental)
  Interventions: Other: Effect of Protein on Blastocyst Development
- 5 mg/ml protein concentration in Embryo Culture Media (No Intervention)

INTERVENTIONS:
Other: Effect of Protein on Blastocyst Development — Embryo Development Related to The Protein Concentration
  Arms: 10 mg/ml protein concentration in Embryo Culture Media

SUMMARY:
Protein Concentration in Human Embryo Culture Media remains assigned to the manufacturers with no clear evidence on which concentration is ideal.

ELIGIBILITY:
Inclusion Criteria:

* Intracytoplasmic sperm injection cycles

Exclusion Criteria:

-

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 1536 (Actual)
Dates: Start 2018-08-14 (Actual); Primary Completion 2020-03-02 (Actual); Study Completion 2020-03-02 (Actual)

PRIMARY OUTCOMES:
Ongoing pregnancy rate | 12 weeks

SECONDARY OUTCOMES:
embryo development | two months
Blastocyst Formation | two months
  number of formed blastocyst per fertilized oocyte
Clinical pregnancy rate | 7 weeks
Implantation rate | 7 weeks
Miscarriage rate | 12 weeks

CONTACTS AND LOCATIONS:
Locations (2):
- Egypt (2):
  - Banon Assiut, Asyut
  - IbnSina IVF Center, Sohag

IPD SHARING:
Plan to Share IPD: No